CLINICAL TRIAL: NCT06854419
Title: Efficacy Evaluation of Blood Peach Extract and Rose Apple Extract on Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CMUH114-REC3-005
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Dermatology
Keywords: skin analysis; skin care products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Drink
- Blood Peach Extract (Experimental)
  Interventions: Dietary Supplement: Blood Peach Extract Drink
- Rose Apple Extract (Experimental)
  Interventions: Dietary Supplement: Rose Apple Extract Drink

INTERVENTIONS:
Dietary Supplement: Placebo Drink — Take one bottle of the product every morning on an empty stomach
  Arms: Placebo
Dietary Supplement: Blood Peach Extract Drink — Take one bottle of the product every morning on an empty stomach
  Arms: Blood Peach Extract
Dietary Supplement: Rose Apple Extract Drink — Take one bottle of the product every morning on an empty stomach
  Arms: Rose Apple Extract

SUMMARY:
Evaluate the effects of blood peach extract drink and rose apple extract drink on enhancing hemoglobin and iron levels, and improving skin health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult females aged 20 to 65;
* Preferably those with pale complexion or signs of iron deficiency anemia.

Exclusion Criteria:

* Currently undergoing or having undergone any medical beauty treatments within the past month (including skincare, laser treatments, chemical peel, injections, or cosmetic surgery);
* Outdoor workers (exposed to sunlight for more than 5 hours daily);
* Pregnant, breastfeeding, or planning to become pregnant during the trial (self-reported);
* Individuals with heart, liver, kidney, endocrine, or other significant organic diseases (self-reported);
* Individuals who have undergone major surgery (according to medical history);
* Long-term medication users;
* Individuals with mental health disorders;
* Those who are already regularly taking iron supplements;
* Faculty or staff members who are currently enrolled in the principal investigator's courses.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
the volume of skin wrinkles | Volume change from Baseline skin wrinkles at 8 weeks
  IRV full-face skin analyzer was utilized to measure skin wrinkles. Units: arbitrary units
the roughness of skin texture | Rating skin roughness from Baseline skin texture at 8 weeks
  IRV full-face skin analyzer was utilized to measure skin texture. Units: arbitrary units

SECONDARY OUTCOMES:
the change of skin elasticity | Change from Baseline skin elasticity at 8 weeks
  Cutometer® was utilized to measure skin elasticity. Units: arbitrary units
the change of skin collagen density | Change from Baseline skin collagen density at 8 weeks
  Dermalab® Combo was utilized to measure skin collagen density. Units: arbitrary units
the change of skin pores | Change from Baseline skin pores at 8 weeks
  IRV full-face skin analyzer was utilized to measure skin pores. Units: arbitrary units
the change of skin tone | Change from Baseline skin tone at 8 weeks
  IRV full-face skin analyzer was utilized to measure skin tone. Units: arbitrary units
the change of skin hydration | Change from Baseline skin hydration at 8 weeks
  Corneometer® was utilized to measure skin hydration. Units: arbitrary units
the change of skin melanin/erythema index | Change from Baseline skin melanin/erythema index at 8 weeks
  Mexameter® was utilized to measure skin melanin/erythema index. Units: arbitrary units
the change of skin redness | Change from Baseline skin redness at 8 weeks
  Colorimeter was utilized to measure skin redness. Units: arbitrary units
the change of lip redness | Change from Baseline lip redness at 8 weeks
  Antera 3D® was utilized to measure lip redness. Units: arbitrary units
the change of Red Blood Cells (RBC) Count of blood | Change from Baseline RBC count at 8 weeks
  venous blood was sampled to measure RBC count
the change of hemoglobin level of blood | Change from Baseline hemoglobin level at 8 weeks
  venous blood was sampled to measure hemoglobin level
the change of mean corpuscular volume (M.C.V) level of blood | Change from Baseline M.C.V level at 8 weeks
  venous blood was sampled to measure M.C.V level
the change of mean corpuscular hemoglobin concentration (M.C.H.C) level of blood | Change from Baseline M.C.H.C level at 8 weeks
  venous blood was sampled to measure M.C.H.C level
the change of ferrous level of blood | Change from Baseline ferrous level at 8 weeks
  venous blood was sampled to measure ferrous level
the change of ferritin level of blood | Change from Baseline ferritin level at 8 weeks
  venous blood was sampled to measure ferritin level
the change of Total Iron Binding Capacity (TIBC) level of blood | Change from Baseline TIBC level at 8 weeks
  venous blood was sampled to measure TIBC level
the change of unsaturated iron-binding capacity (UIBC) level of blood | Change from Baseline UIBC level at 8 weeks
  venous blood was sampled to measure UIBC level

OTHER OUTCOMES:
the change of liver function biomarkers (AST, ALT) of blood | change from Baseline liver function biomarkers at 8 weeks
  venous blood was sampled to measure liver function biomarkers
the change of renal function biomarkers (creatinine, BUN) of blood | change from Baseline renal function biomarkers at 8 weeks
  venous blood was sampled to measure renal function biomarkers
the change of fasting glucose level of blood | change from Baseline fasting glucose level at 8 weeks
  venous blood was sampled to measure fasting glucose level
the change of Advanced glycation end products (AGEs) level of blood | change from Baseline AGEs level at 8 weeks
  venous blood was sampled to measure AGEs level
The change of self-assessment skin and metabolic circulation condition | Change from Baseline skin and metabolic circulation condition at 8 weeks
  A self-assessment questionnaire was collected to evaluate skin and metabolic circulation condition. As for the evalutation of skin condition, the higher score the better; As for evaluation of metabolic circulation condition, the higher score the worse.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Mei Chiang, Principal Investigator — China Medical University of Department of Cosmeceutics
Locations (1):
- China Medical University of Department of Cosmeceutics, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No